CLINICAL TRIAL: NCT00435422
Title: Neuroaxial Blokade and the Effect of Fluid Optimization
Brief Title: Neuroaxial Blokade and Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Henrik Kehlet, prof., PhD, Rigshospitalet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neuroaxial blokade and BP
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2009-02

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

INTERVENTIONS:
Procedure: Stroke volume optimization — Stroke volume optimization

SUMMARY:
The effect of individualized fluid optimization during neuroaxial blockade has not been evaluated. The investigators evaluated if if Stroke decrease 15 min after activation of neuroaxial blockade and whether SV could be optimized to pre activation values.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate SV maximization with aid of the LiDCO system which is a minimal invasive technique only requiring a venous and arterial line. We thereby attempt to cover the specific individual fluid deficit induced by neuroaxial blockade.

ELIGIBILITY:
Inclusion Criteria:

* Neuroaxial blockade (thoracic)

Exclusion Criteria:

* Weight below 40 kg
* Lithium therapy
* Type I diabetes or type II requiring insulin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Stroke volume | 15 min after blockade

SECONDARY OUTCOMES:
Brain oxygenation, cardiac output, TPR, NIRS, BP | 15 min after blockade

CONTACTS AND LOCATIONS:
Overall Officials: Morten Bundgaard-Nielsen, MD, Principal Investigator — Section of surgical pathophysiology; Morten Bundgaard-Nielsen, MD, Principal Investigator — unafiliated
Locations (1):
- Rigshospitalet, Copenhagen, Denmark